CLINICAL TRIAL: NCT00825838
Title: A Randomized Double-Blind Placebo-Controlled Clinical Trial of a Purified Chili Pepper Extract (CH-19 Sweet Extract) to Evaluate Its Safety and Efficacy for Weight and Fat Loss and Metabolism Change in Overweight or Obese Healthy Male and Female Adults
Brief Title: Effect of Chili Pepper Extract on Weight and Fat Loss and Metabolism Increase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ajinomoto USA, INC. (Industry)
Responsible Party: Kentaro Maruyama, Ajinomoto USA, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CH19-001
Record Dates: First submitted 2009-01-18; First posted 2009-01-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Overweight; Obesity
Keywords: Body weight; Body composition; Resting metabolic rate and fat oxidation in men; class I obese
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Oral ingestion of 6mg chili pepper extract
  Interventions: Dietary Supplement: Chronic consumption of chili pepper extract
- 2 (Placebo Comparator): Oral ingestion of 0 mg chili pepper extract (matching placebo)
  Interventions: Dietary Supplement: Chronic consumption of matching placebo

INTERVENTIONS:
Dietary Supplement: Chronic consumption of chili pepper extract — 6mg chili pepper extract per day in two divided doses (before the morning meal and before the evening meal) up to 12 weeks.
  Arms: 1
Dietary Supplement: Chronic consumption of matching placebo — 0mg chili pepper extract (matching placebo) per day in two divided doses (before the morning meal and before the evening meal) up to 12 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to test the safety and effectiveness of a purified extract of CH-19 Sweet, containing capsinoids.

ELIGIBILITY:
Inclusion Criteria:

* Is overweight or obese but otherwise generally healthy who interested in losing weight
* BMI of 25 to 35 kg/m2
* Waist/hip ratio of 0.9 or more for male and 0.85 for female.

Exclusion Criteria:

* Type 1 or 2 diabetes mellitus
* cardiovascular disease (other than mild, controlled hypertension or dislidemia)
* On a weight-loss program within six months

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2006-04; Primary Completion 2006-10 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
body weight and body composition | 12 weeks

SECONDARY OUTCOMES:
resting metabolic rate and substrate oxidation | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soren Snitker, M.D., Ph.D., Study Chair — University of Maryland, Baltimore; Yoshiyuki Fujishima, D. Phil., Study Director — Ajinomoto USA, INC.